CLINICAL TRIAL: NCT06239467
Title: PIKture-01: First-in-Human Study of the PI3KαH1047R Mutant-Selective Inhibitor OKI-219 as Monotherapy in Participants With Advanced Solid Tumors and as Part of Combination Therapy in Participants With Advanced Breast Cancer
Brief Title: First-in-Human Study of OKI-219 in Advanced Solid Tumors and Advanced Breast Cancer
Acronym: PIKture-01
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: OnKure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OKI-219-101
Record Dates: First submitted 2024-01-12; First posted 2024-02-02 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Advanced Cancer; Breast Cancer; Advanced Solid Tumors; PI3K Gene Mutation
Keywords: PI3K; Solid Tumor; Breast Cancer; OKI-219; trastuzumab; fulvestrant; H1047r; ribociclib; atirmociclib; tucatinib
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; Trastuzumab; tucatinib; ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Phase 1a: Part A Dose Escalation (Experimental): OKI-219 Monotherapy Dose Escalation in participants with advanced solid tumors with the PI3KαH1047R mutation
  Interventions: Drug: OKI-219
- Phase 1b: Part B Dose Escalation (Experimental): OKI-219 + Fulvestrant Dose Escalation in participants with HR+/HER2- locally advanced, unresectable or metastatic breast cancer with the PI3KαH1047R mutation
  Interventions: Drug: OKI-219; Drug: Fulvestrant
- Phase 1b: Part B Dose Optimization (Experimental): OKI-219 + Fulvestrant Dose Optimization in participants with HR+/HER2- locally advanced, unresectable or metastatic breast cancer with the PI3KαH1047R mutation
  Interventions: Drug: OKI-219; Drug: Fulvestrant
- Phase 1b: Part C Dose Escalation (Experimental): OKI-219 + Tucatinib + Trastuzumab Dose Escalation in participants with HR±/HER2+ locally advanced, unresectable or metastatic breast cancer with the PI3KαH1047R mutation
  Interventions: Drug: OKI-219; Drug: Trastuzumab; Drug: Tucatinib
- Phase 1b: Part C Dose Expansion (Experimental): OKI-219 + Tucatinib + Trastuzumab Dose Expansion in participants with HR±/HER2+ locally advanced, unresectable or metastatic breast cancer with the PI3KαH1047R mutation
  Interventions: Drug: OKI-219; Drug: Trastuzumab; Drug: Tucatinib
- Phase 1b: Part D Dose Escalation (Experimental): OKI-219 + Fulvestrant + Atirmociclib Dose Escalation in participants with HR+/HER2- locally advanced, unresectable or metastatic breast cancer with the PI3KαH1047R mutation
  Interventions: Drug: OKI-219; Drug: Fulvestrant; Drug: Atirmociclib
- Phase 1b: Part D Dose Expansion (Experimental): OKI-219 + Fulvestrant + Atirmociclib Dose Escalation in participants with HR+/HER2- locally advanced, unresectable or metastatic breast cancer with the PI3KαH1047R mutation
  Interventions: Drug: OKI-219; Drug: Fulvestrant; Drug: Atirmociclib
- Phase 1b: Part E Dose Escalation (Experimental): OKI-219 + Fulvestrant + Ribociclib Dose Escalation in participants with HR+/HER2- locally advanced, unresectable or metastatic breast cancer with the PI3KαH1047R mutation
  Interventions: Drug: OKI-219; Drug: Fulvestrant; Drug: Ribociclib
- Phase 1b: Part E Dose Expansion (Experimental): OKI-219 + Fulvestrant + Ribociclib Dose Expansion in participants with HR+/HER2- locally advanced, unresectable or metastatic breast cancer with the PI3KαH1047R mutation
  Interventions: Drug: OKI-219; Drug: Fulvestrant; Drug: Ribociclib

INTERVENTIONS:
Drug: OKI-219 — Oral twice daily
Drug: Fulvestrant — Intramuscular injection
  Arms: Phase 1b: Part B Dose Escalation; Phase 1b: Part B Dose Optimization; Phase 1b: Part D Dose Escalation; Phase 1b: Part D Dose Expansion; Phase 1b: Part E Dose Escalation; Phase 1b: Part E Dose Expansion
Drug: Trastuzumab — Intravenous (IV)
  Arms: Phase 1b: Part C Dose Escalation; Phase 1b: Part C Dose Expansion
Drug: Tucatinib — Oral twice daily
  Arms: Phase 1b: Part C Dose Escalation; Phase 1b: Part C Dose Expansion
Drug: Atirmociclib — Oral twice daily
  Arms: Phase 1b: Part D Dose Escalation; Phase 1b: Part D Dose Expansion
Drug: Ribociclib — Oral once daily continuous for 21-days followed by 7 days off
  Arms: Phase 1b: Part E Dose Escalation; Phase 1b: Part E Dose Expansion

SUMMARY:
OKI-219-101 is a Phase 1a/1b, open-label, multicenter, dose-escalation study designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PDx), and efficacy of OKI-219 as monotherapy and in combination with other anti-cancer drugs. Phase 1a (Part A) will investigate escalating doses of OKI-219 monotherapy, and Phase 1b will investigate OKI-219 (at a tolerated dose determined in Part A) in combination with fulvestrant (Part B), trastuzumab and tucatinib (Part C), atirmociclib (Part D), and ribociclib and fulvestrant (Part E). Participants will continue to receive study treatment until disease progression, intolerable toxicity, or other study treatment withdrawal criteria are met.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with advanced solid tumors with documented evidence of a PI3KαH1047R mutation in tumor tissue and/or blood (ie, ctDNA).
* Eastern Cooperative Oncology Group (ECOG) Performance status score of to 1.
* Life expectancy > 12 weeks for Part A and > 6 months for Parts B, C, D, and E in the opinion of the Investigator.
* Adequate organ and bone marrow function
* Have adequate archival tumor tissue sample available or be approved by the Sponsor for enrollment if no tumor sample is available.
* At least 1 measurable lesion based on RECIST version 1.1.

Additional Cohort-specific key inclusion criteria:

Part A

* Participants with HR+/HER2- locally advanced, unresectable or metastatic breast cancer, must have received at least 1 prior line of hormonal therapy and at least 1 prior line of CDK4/6-inhibitor in the advanced or metastatic setting.
* Participants with HER2+ locally advanced, unresectable or metastatic breast cancer, must have received prior taxane, trastuzumab, pertuzumab, and tucatinib. Prior trastuzumab deruxtecan is allowed but not required.
* Participants with HER2-low breast cancer must have received prior trastuzumab deruxtecan.
* Participants with colorectal cancer must have KRAS wild-type disease.

Part B

* Participants with locally advanced, unresectable or metastatic HR+/HER2- breast cancer must have received at least 1 prior line of hormonal therapy in the advanced or metastatic setting and at least 1 prior CDK4/6-inhibitor.
* Participants with HER2-low breast cancer should have received prior trastuzumab deruxtecan

Part C ● Participants with HR±/HER2+ locally advanced, unresectable or metastatic breast cancer must have received prior taxane, trastuzumab, and pertuzumab unless unavailable in the region or contraindicated. Prior trastuzumab deruxtecan is allowed but not required.

Part D

● Participants must have HR+/HER2- locally advanced, unresectable or metastatic breast cancer

Part E ● Participants must have HR+/HER2- locally advanced, unresectable or metastatic breast cancer.

Key Exclusion Criteria:

* Treatment with any investigational product or other anticancer therapy within 28 days or 5 half-lives, whichever is shorter, of the start of treatment
* Participants with a known KRAS mutation.
* Participants with a known deleterious mutation in phosphatase and tensin homolog (PTEN) or negative for PTEN protein expression by IHC.
* Major surgery or wide-field radiation within 28 days or limited field palliative radiation within 7 days prior to the first dose of study drug.
* Known active central nervous system metastasis, including leptomeningeal disease.
* Uncontrolled Type 1 or Type 2 diabetes as defined by HbA1C ≥ 8%.
* Concomitant active malignancy or previous malignancy within 2 years of the time of enrollment.
* Impaired cardiovascular function or clinically significant cardiovascular disease,
* History of symptomatic drug-induced pneumonitis.
* Participants with active HIV, Hepatitis B, and Hepatitis C viral infections

Additional Cohort-specific key exclusion criteria:

Part C:

* Grade 2 or higher diarrhea at study entry.
* History of chronic liver disease.

Part E:

● History of interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Identify maximum tolerated dose (MTD) of OKI-219 in monotherapy | Cycle 1 (First 28 days on treatment)
  Frequency of participants experiencing dose-limiting toxicities during the first 28-day cycle
Assess safety of OKI-219 as monotherapy or in combination with other anti-cancer therapies: incidence of SAEs | Through 30 days after last dose, an average of 1 year
  Number and type of SAEs experienced by participants during treatment and follow-up
Assess safety of OKI-219 as monotherapy or in combination with other anti-cancer therapies: incidence of Grade 2 or greater treatment emergent adverse events | Through 30 days after last dose, an average of 1 year
  Number of treatment-emergent adverse events (TEAEs) equal or greater than Grade 2 experienced during treatment and follow-up
Assess rate of dose modifications during treatment with OKI-219 as monotherapy or in combination with other anti-cancer therapies | Through last study dose, an average of 1 year
  rate of dose modifications

SECONDARY OUTCOMES:
Assess the plasma PK of OKI-219 following single and multiple doses as monotherapy or in combination with other anti-cancer therapies: maximum plasma concentration (Cmax) | Through cycle 6 of treatment (up to 28 weeks)
  PK of OKI-219: Cmax
Assess the plasma PK of OKI-219 following single and multiple doses as monotherapy or in combination with other anti-cancer therapies: time of maximum plasma concentration (Tmax) | Through cycle 6 of treatment (up to 28 weeks)
  PK of OKI-219: Tmax
Assess the plasma PK of OKI-219 following single and multiple doses as monotherapy or in combination with other anti-cancer therapies: area under the plasma concentration-time curve (AUC) | Through cycle 6 of treatment (up to 28 weeks)
  PK of OKI-219: AUC
Assess the plasma PK of OKI-219 following single and multiple doses as monotherapy or in combination with other anti-cancer therapies: terminal elimination half-life time (t1/2) | Through cycle 6 of treatment (up to 28 weeks)
  PK of OKI-219: t1/2
To estimate the preliminary antitumor activity of OKI-219 as monotherapy and in combination with other anti-cancer therapies: objective response rate (ORR) | Up to approximately 36 months
  ORR per investigator assessed Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1)
To estimate the preliminary antitumor activity of OKI-219 as monotherapy and in combination with other anti-cancer therapies: clinical benefit rate (CBR) | Up to approximately 36 months
  CBR per investigator assessed Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1)
Dose optimization only: to estimate the preliminary antitumor activity of OKI-219 as monotherapy and in combination with other anti-cancer therapies: progression free survival (PFS) | Up to approximately 36 months
  PFS per investigator assessed Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1)
To assess the dose-response impact of OKI-219 as monotherapy and in combination with other anti-cancer therapies on PI3KαH1047R ctDNA levels | Through last study dose, an average of 1 year
  Changes in PI3KαH1047R ctDNA on treatment and end of treatment (EOT) compared to baseline.
To determine the impact of OKI-219 dosing as monotherapy and in combination with other anti-cancer therapies on blood glucose and insulin | Through last study dose, an average of 1 year
  Changes in plasma glucose, serum insulin, serum c-peptide levels, and hemoglobin A1c (HbA1c) will be evaluated on treatment compared to baseline.
To assess the PDx activity of OKI-219 as monotherapy and in combination with other anti-cancer therapies | Through last study dose, an average of 1 year
  PDx activity will be evaluated with serial tumor biopsy samples assessed for PI3K/AKT/mTOR downstream pathway changes.

CONTACTS AND LOCATIONS:
Locations (34):
- United States (13):
  - California Cancer Associates for Research and Excellence, Encinitas, California
  - University of California San Diego UCSD, La Jolla, California
  - UCLA Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Hoag - Huntington Beach, Newport Beach, California
  - Regents of the University of Colorado, Aurora, Colorado
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Insitute, Detroit, Michigan
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Stony Brook University, Stony Brook, New York
  - SCRI Oncology Partners - Nashville, Nashville, Tennessee
  - NEXT Oncology Virginia, Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Belgium (3):
  - Institut Jules Bordet, Anderlecht
  - UZ Leuven - Campus Gasthuisberg, Leuven
  - GZA Hopsitals Campus Sint-Augustinus, Wilrijk
- France (6):
  - Centre de Lutte Contre le Cancer CLCC - Centre Georges Francois Leclerc (CGFL), Dijon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Centre Antoine Lacassagne, Nice
  - Hopital Lyon Sud, Pierre-Bénite
  - Institut Gustave Roussy, Villejuif
- Italy (3):
  - Ospedale San Raffaele, Milan
  - Ospedale San Gerardo-ASST Monza, Monza
  - Istituto Clinico Humanitas, Rozzano
- South Korea (5):
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (4):
  - NEXT Oncology Phase I Unit / IOB- Hospital Quironsalud Barcelona, Barcelona
  - Hospital Beata Maria Ana, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - START - Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No